CLINICAL TRIAL: NCT04306757
Title: Flow Controlled Ventilation Versus Pressure Controlled Ventilation in Cardiac Surgery After Cardiopulmonary Bypass Without Ventilation - a Prospective, Randomized Clinical Study
Brief Title: Flow Controlled Ventilation in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1211/2019
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Respiration; Artificial; Positive-Pressure Respiration
Keywords: flow controlled ventilation; pressure controlled ventilation; cardiac surgery
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: controlled, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCV (Experimental): Artificial ventilation will be performed with individualized flow-controlled ventilation (Evone, Ventinova Medical B.V., Eindhoven, the Netherlands) during cardiac surgery until admission to postoperative ICU. Individualisation will be established by compliance guided end-expiratory and peak pressure setting, flow setting will be adjusted to secure normocapnia and I:E Ratio set to 1:1.
  Interventions: Device: Evone
- PCV (Active Comparator): Artificial ventilation will be performed with low tidal volume pressure-controlled ventilation (Primus, Dräger, Lübeck, Germany) during cardiac surgery until admission to postoperative ICU. Peak pressure will be set to achieve a tidal volume of 7ml/kg predicted body weight at a compliance titrated positive end-expiratory pressure. Respiratory rate will be set to maintain normocapnia and I:E ratio set to 1:1.5 except extension of expiration is necessary in order to avoid air trapping.
  Interventions: Device: Primus

INTERVENTIONS:
Device: Evone — Airway ventilation device
  Arms: FCV
Device: Primus — Airway ventilation device
  Arms: PCV

SUMMARY:
This trial investigates effects of individualized (by compliance guided pressure settings) flow-controlled ventilation compared to best clinical practice pressure controlled ventilation in cardiac surgery requiring cardiopulmonary bypass.

DETAILED DESCRIPTION:
The aim of the study is to investigate flow-controlled ventilation (FCV) during cardiac surgery requiring cardiopulmonary bypass. Previous preclinical trials have already shown improved oxygenation and CO2 removal within a significantly reduced respiratory minute volume as an expression of more efficient gas exchange with FCV compared to volume controlled ventilation (VCV). Preliminary data of our own animal study comparing individualized FCV by compliance guided pressure settings with state-of-the-art low tidal volume pressure controlled ventilation (PCV) confirmed previous findings with a significantly improved oxygenation by 20% while reducing respiratory minute volume. We therefore assume that FCV may be a more lung protective ventilation method.

Open heart surgery requires bridging of the heart and lung function with a cardiopulmonary bypass (CPB) performed by a heart-lung machine. During this time the lung is most frequently not ventilated at all and lies collapsed in the chest for several hours. After weaning from CPB, the lungs must be recruited and ensure sufficient gas exchange of the blood. Not surprisingly, the incidence of postoperative pulmonary complications (PPC) at 20-30% is comparatively high after cardiac surgery and is the leading cause of perioperative mortality. Based on previous trials we expect improved oxygenation and thus arterial partial pressure of oxygen (pO2) is the main primary outcome parameter of this study. Furthermore, we expect improved recruitment of lung tissue due to controlled expiratory flow in FCV without the need of recruitment maneuvers, which may cause deleterious effects on lung tissue. Thus, lung tissue aeration assessed by Hounsfield units analyses of a postoperative computed tomography will be a secondary outcome parameter.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects >18 years
* Body weight >40 kg
* Elective cardiac surgery with CPB and without ventilation during CPB
* American Society of Anaesthesiologists (ASA) risc classification I-IV
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Female subjects known to be pregnant
* Known participation in another interventional clinical trial
* High risk cardiac surgery such as double valve surgery, re-cardiac surgery, intraoperative cardiac arrest or pre-existing high grade cardiomyopathy (ejection fraction <30%)
* Closing operation field without chest closure due to hemodynamic instability
* Acute endocarditis under antibiotic treatment
* Minimal invasive valve surgery via thoracotomy (MIC)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Horowitz Index | 15 minutes after chest closure
  arterial partial pressure of Oxygen (paO2) / fraction of inspired Oxygen (FiO2)

SECONDARY OUTCOMES:
lung tissue aeration | immediately postoperative
  Lung tissue aeration assessed by Hounsfield units analysis of computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Judith Martini, MD, Principal Investigator — Medical University Innsbruck, Dept. of Anaesthesiology
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt J, Wenzel C, Mahn M, Spassov S, Cristina Schmitz H, Borgmann S, Lin Z, Haberstroh J, Meckel S, Eiden S, Wirth S, Buerkle H, Schumann S. Improved lung recruitment and oxygenation during mandatory ventilation with a new expiratory ventilation assistance device: A controlled interventional trial in healthy pigs. Eur J Anaesthesiol. 2018 Oct;35(10):736-744. doi: 10.1097/EJA.0000000000000819. PMID 29734208